CLINICAL TRIAL: NCT07211607
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous Selonabant in Healthy Adult Subjects Aged 18 to 30 Years
Brief Title: I.V. Selonabant in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anebulo Pharmaceuticals (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-IV-25-01
Record Dates: First submitted 2025-09-29; First posted 2025-10-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: single ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Experimental Cohort 1 (Experimental): Single intravenous dose of 1 mg of selonabant or placebo
  Interventions: Drug: selonabant; Drug: placebo
- Experimental Cohort 2 (Experimental): Single intravenous dose of 2 mg of selonabant or placebo
  Interventions: Drug: selonabant; Drug: placebo
- Experimental Cohort 3 (Experimental): Single intravenous dose of 5 mg of selonabant or placebo
  Interventions: Drug: selonabant; Drug: placebo
- Experimental Cohort 4 (Experimental): Single intravenous dose of 10 mg of selonabant or placebo
  Interventions: Drug: selonabant; Drug: placebo
- Experimental Cohort 5 (Experimental): Single intravenous dose of 20 mg of selonabant or placebo
  Interventions: Drug: selonabant; Drug: placebo

INTERVENTIONS:
Drug: selonabant — Intravenous infusion of selonabant
  Other Names: ANEB-001
Drug: placebo — Placebo infusion which looks the same as the selonabant infusion

SUMMARY:
This is a Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous Selonabant in Healthy Adult Subjects Aged 18 to 30 Years

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, SAD study to evaluate the safety, tolerability, and PK of single IV doses of selonabant in healthy adult participants between 18 and 25 years of age. The study will enroll up to 5 sequential cohorts of 8 subjects (6 active, 2 placebo) for a total of up to 40 subjects. The starting dose of selonabant will be 1 mg and the planned doses for subsequent cohorts are 2, 5, 10, and 20 mg. The study is supported by a collaborative U01 grant from NIDA.

ELIGIBILITY:
Key Inclusion Criteria:

1. The subject is male or female 18 to 30 years of age, inclusive.
2. The subject has a body mass index of 18 to 30 kg/m2, inclusive, and with a minimum weight of 50 kg and maximum weight of 110 kg.
3. The subject has no clinically significant medical history and no clinically significant findings in vital sign measurements, 12-lead ECG results, and physical examination findings at screening that would pose a risk in study participation, as determined by the investigator. The subject has no clinical laboratory test results outside the reference range that remain out of range after up to 2 repeat tests within the screening window.
4. The female subjects must be surgically sterile (ie, hysterectomy and/or oophorectomy) or agree to use a highly effective method of birth control in addition to a secondary barrier method of contraception during the study and for at least 110 days (90 days plus 5 selonabant half-lives, assuming a half-life of 80 hours) after dosing with study treatment.

Key Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject has used any prescription (excluding hormonal birth control) or over the counter medications within 14 days or less than 5 half-lives (whichever is longer) of screening and for the entire duration of the study. Exceptions will only be made upon the investigator's decision and discussion with the Sponsor.
3. The subject has used any vitamin, mineral, herbal, or dietary supplements within 14 days or less than 5 half-lives (whichever is longer) of screening and for the entire duration of the study. Exceptions will only be made upon the investigator's decision and discussion with the Sponsor.
4. The subject has used any cannabis products within 14 days of study drug administration.
5. The subject uses any anti-anxiety, anti-depressant, anti-psychotic, anti-epileptic, or anti-migraine medication.
6. The subject has a positive urine drug screen result for drugs of abuse at screening or check-in.
7. The subject has a history of alcohol abuse or drug addiction within the last year
8. The subject's alcohol urine test at screening or check-in was positive. Alcohol will not be allowed for at least 24 hours before screening or check-in until discharge.
9. The subject has used nicotine- or tobacco-containing products in the last 3 months. Smoking and nicotine use will not be allowed during the study.
10. The subject has used any caffeine-containing food or drink (eg, tea, coffee, cola, chocolate) or 'energy' drinks within 24 hours before study admission. Caffeine containing food and drink will not be allowed from at least 24 hours before screening or check-in until discharge.
11. The subject has received a diagnosis (or tests positive at screening) for hepatitis B or hepatitis C.
12. The subject has a history of HIV, or tests positive for HIV, or has evidence of active tuberculosis (history and/or radiology findings) at screening.
13. The subject has a medical history of impaired cardiac function or clinically significant cardiac disease
14. The subject has an estimated glomerular filtration rate of <90 mL/min/1.73 m2, based on the CKD-EPI equation.
15. The subject has any abnormal, out-of-range screening laboratory values that remain outside laboratory-defined limits after up to 2 repeat tests within the screening window.
16. The subject has SBP >130 or <90 mm Hg, and DBP >95 or <50 mm Hg at screening or check-in. If a subject fails to meet SBP and/or DBP criteria, up to 2 repeat measurements, one via automated device and one via manual reading, may be completed after the subject has remained in the seated position for 5 minutes between readings, at the discretion of the investigator. For those subjects who have a repeat blood pressure measurement, the repeat value will be used to determine eligibility.
17. The subject had a loss of blood or donated blood or blood products >500 mL within 4 months prior to screening or has the intention to donate blood or blood products during the study.
18. The subject has a baseline coagulation test result outside the normal range for the clinical site.
19. The subject has a history of arterial or venous thrombosis or a family history of a coagulopathy.
20. The subject has any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as a history of seizures (excluding febrile convulsions below 3 years of age).
21. The subject has a current psychiatric disorder (including depression), schizophrenia, bipolar disorders, eating disorders, personality disorders, post-traumatic stress disorders, anxiety disorders (including panic, obsessive-compulsive disorders, and phobias), a history of depression or suicidal ideation, or a history of suicide attempt.
22. The subject has a current or history of neurological disease, including but not limited to, seizure disorder, cerebrovascular disease, intractable headache syndromes (e.g. intractable migraines, history of eclampsia, cluster headaches), multiple sclerosis, ataxias, and extrapyramidal disorders.
23. The subject has a positive test for SARS-CoV-2.
24. The subject has a history of serious hypersensitivity reaction to a known ingredient of selonabant or excipients.
25. The subject has received study drug (selonabant) in any investigational study or received any other investigational study drug in any other study within 30 days of dosing or 5 half lives, whichever is longer.
26. The subject has difficult venous access or a history of infusion site reactions, including local tissue reactions, hyperpyrexia, or any related reactions.
27. The subject has intercurrent illness that is either life threatening or of clinical significance such that it might limit compliance with study requirements, or in the investigator's assessment would place the subject at an unacceptable risk for study participation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 28 days
Number of Participants with Clinically Significant Laboratory Test Results | 28 days
Number of Participants with Clinically Significant Vital Signs Values | 28 days
Number of Participants with Clinically Significant Abnormal ECG Findings | 28 days
Number of Participants with Clinically Significant Abnormal Physical Exam Findings | 28 days
Change from Baseline in Beck Depression Inventory (BDI) | 28 days
  The minimum possible Beck Depression Inventory (BDI) score is 0, and the maximum score is 63. This score is determined by summing the ratings from the 21 questions, with each question scoring from 0 to 3, indicating the severity of depressive symptoms over the past two weeks. Lower score means less depression
Change from Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) | 28 days
  The Columbia-Suicide Severity Rating Scale (C-SSRS) does not have a single minimum or maximum score, as it is not a traditional cumulative-score test. Instead, it uses a series of "yes" or "no" questions to place an individual into distinct categories of risk based on their specific responses. Lower score means less suicidal ideation.
Area Under the Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration | 28 days
Terminal Elimination Phase Half-life (T1/2) | 28 days
Maximum Observed Concentration (Cmax) | 28 days
Pharmacokinetic Clearance (CL) | 28 days
  Pharmacokinetic clearance (\(CL\)) is a quantitative measure of how efficiently the body removes a drug from the bloodstream. It is defined as the volume of plasma from which a drug is completely and irreversibly removed per unit of time and is typically expressed in units like milliliters per minute (mL/min) or liters per hour (L/h).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Gilbey, MD, Principal Investigator — PPD Austin Clinical Research Unit; Rebecca Wood-Horrall, MD, Study Chair — PPD Austin Clinical Research Unit
Locations (1):
- PPD Austin Clinical Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No